CLINICAL TRIAL: NCT06601868
Title: The Impact of Nutritional Optimization to Enhance Postoperative Outcomes Using the R-Support Supplements
Acronym: R-Support
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: Chirec (Other); Zuyderland Medical Centre (Other)
Responsible Party: Principal Investigator, Letizia Georgiou, Research Fellow in Plastic Surgery, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23440_R-Support
Record Dates: First submitted 2024-08-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Abdominoplasty; Breast Reduction; Autologous Breast Reconstruction; Body Contouring Surgery

STUDY DESIGN:
Intervention Model Description: This pilot study will include a total of 200 patients. Participants will be randomly assigned to one of two groups using a randomization algorithm. The study will be non-blinded, meaning both participants and researchers will be aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 100 patients without R-Support supplementation (control group) (No Intervention): These patients will have no intervention, will not take the nutritional supplements
- 100 patients with R-Support supplementation (intervention group) (Active Comparator): The treatment period for the intervention group will last 28 days, divided into two phases: 14 days preoperative and 14 days postoperative.
  During the preoperative phase, participants will consume one shake per day. Each shake will consist of 35 grams (3 scoops) of R-Support Prepare mixed with 250 milliliters of water or milk. This regimen will be followed for 14 days leading up to the surgery.
  During the postoperative phase, participants will consume one shake per day. Each shake will consist of 35 grams (3 scoops) of R-Support After mixed with 250 milliliters of water or milk. This regimen will be followed for 14 days following the surgery.
  Interventions: Dietary Supplement: R-Support Prepare & After nutritional supplement

INTERVENTIONS:
Dietary Supplement: R-Support Prepare & After nutritional supplement — R-Support is a nutritional supplement containing proteins, Vitamine A, Vitamine B6, Vitamine B11, Vitamine B12, Vitamine C, Vitamine D3, Vitamine E, IJzer, Koper, Selenium, Zink, Magnesium, Omega-3 and Beta-glucanen.
  Arms: 100 patients with R-Support supplementation (intervention group)

SUMMARY:
The aim of this pilot study is to evaluate the potential benefits of nutrient supplementation on post-operative recovery for patients undergoing certain types of surgery, compared to those who do not receive such supplementation. The multi-center study will be conducted in Belgium and the Netherlands at UZ Brussel, Delta CHIREC, and Zuyderland Medical Center.

The pilot study will serve as a precursor to a randomized controlled trial and will include 200 patients. Participants must be classified as ASA I or II, aged between 18 and 65, and undergoing abdominoplasty, breast reduction, breast reconstruction through a DIEP-flap, or extensive circumferential liposuction and body contouring surgery.

Eligible patients who provide informed consent will be randomly assigned to either the intervention group, receiving R-Support supplementation, or the control group, without supplementation. Each group will consist of 100 patients. The study will span 8 weeks, with a 2-week preoperative period and a 6-week postoperative period. The treatment will involve a 28-day supplementation period, with R-Support Recover Prepare given 14 days preoperatively and R-Support Recover After given 14 days postoperatively.

Postoperative recovery will be assessed using the PRP-Questionnaire and Functional Recovery Index, which together will measure physical and psychological recovery, as well as the speed of recovery in the early postoperative phase. The study hypothesizes that the intervention group will experience quicker recovery than the control group. Additionally, data on hospital stay duration and early postoperative complications will be collected, with the expectation that better-prepared bodies will recover faster, potentially leading to fewer hospitalized days and complications. The study aims to demonstrate enhanced postoperative recovery, reduced early complications (such as wound dehiscence and infection), and shorter hospital stays.

DETAILED DESCRIPTION:
The aim of this pilot study is to assess the potential for enhanced postoperative recovery in patients receiving nutrient supplementation (intervention) before and after surgery, compared to patients who do not receive nutrient supplementation (control). This is a multi-center study taking place in Belgium and the Netherlands, with study sites including the following hospitals: UZ Brussel (BE), Delta CHIREC (BE), and Zuyderland Medical Center (NL).

This is a pilot study, with the end goal being a randomized controlled trial. A total of 200 patients will be included. The inclusion criteria are participants classified as ASA I or II, aged between 18 and 65, and undergoing one of the following types of surgery: abdominoplasty, breast reduction, breast reconstruction via DIEP-flap, or extensive circumferential liposuction and body contouring surgery.

Every patient who meets the inclusion criteria and provides informed consent will be randomly allocated to either the intervention or control group via a randomization algorithm: 100 patients without R-Support supplementation (control group) and 100 patients with R-Support supplementation (intervention group).

The study will last a total of 8 weeks, divided into a 2-week preoperative period and a 6-week postoperative period. The treatment period will be 28 days: 14 days preoperatively (supplementation with R-Support Recover Prepare) and 14 days postoperatively (supplementation with R-Support Recover After).

Data regarding postoperative recovery will be assessed using the PRP-Questionnaire and the Functional Recovery Index. These two questionnaires combined will provide a comprehensive overview of postoperative recovery, both physically and psychologically, as well as the speed of recovery in the early postoperative phase. The investigators hypothesize that the intervention group (with R-Support) will experience quicker postoperative recovery than the control group (without R-Support). Additionally, data on the length of hospital stay and early postoperative complications (minor, not requiring surgery, such as wound dehiscence <2 cm and localized infection; and major, requiring surgery, such as wound dehiscence >2 cm and infection requiring surgical debridement) will be collected. The investigators suggest that a body better prepared for surgery may, hypothetically, recover more quickly. This could be reflected in fewer hospitalized days and fewer wound complications. The study's endpoints are enhanced postoperative recovery, reduced early complications (wound dehiscence, infection), and shortened hospital stays.

ELIGIBILITY:
Inclusion Criteria:

* ASAI&II
* Age 18-65
* Type of surgery:

  * Abdominoplasty o Breast reduction
  * Breast reconstruction through a DIEaP-flap
  * Extensive circumferential liposuction and body contouring surgery

Exclusion Criteria:

* Patients with systemic illness, including:

  * Diabetes
  * Immune deficiencies
  * Severe cardiovascular disease
  * Renal insufficiency
* Active smokers or smokers that didn't quit 4 weeks prior to surgery
* Patients under chemotherapy (Patients currently undergoing chemotherapy are not allowed to participate in this study. Patient undergoing previous chemotherapy are allowed to participate in this study, as long as the chemotherapy ended 6 months before the planned surgery and are currently in remission or free of disease.)
* Patients after bariatric surgery with partial or complete stomachresection
* Patients taking SSRI medication
* Pregnancy
* ASAIII&IV
* Gluten intolerance
* Lactose intolerance
* Allergy or hypersensitivity to fish, soya, milk, shellfish.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative outcomes assessment: The Functional Recovery Index Questionnaire evaluates pain, social, lower limb, and physical activity, and the Postoperative Recovery Profile assesses physical, psychological, and social factors. | 2 weeks postoperative
  The Functional Recovery Index (FRI) focuses on pain and social activity, with a particular emphasis on lower limb mobility, which is often compromised after surgery. This tool aims to assess whether R-Support supplementation improves mobility and overall recovery.
  Recovery will be quantified using a scale from 0 to 10, where 0 indicates no difficulty at all, and 10 represents extreme difficulty.
Postoperative outcomes assessment: The Postoperative Recovery Profile (PRP) Questionnaire | 6 weeks postoperative
  The Postoperative Recovery Profile (PRP) Questionnaire assesses physical symptoms, functions, psychological aspects, social interactions, and activity levels. Patients will complete both questionnaires independently.
  Recovery will be quantified using a scale from 0 to 10, where 0 indicates no difficulty at all, and 10 represents extreme difficulty. It is hypothesized that patients receiving R-Support will experience a quicker recovery compared to those who do not.

SECONDARY OUTCOMES:
Length of hospital stay | 1 week postoperative
  The postoperative complication assessment will focus on the length of hospital stay, measured in days. This measurement aims to determine whether patients receiving R-Support have a shorter hospital stay compared to those who do not. A reduced length of stay may indicate quicker recovery, highlighting the potential benefits of R-Support supplementation in enhancing postoperative outcomes.
Early postoperative complication assessment | 1 and 2 weeks postoperative
  The early postoperative complication assessment will classify complications into two categories: minor and major.
  Minor complications include issues such as wound dehiscence less than 2 cm and localized infections that do not require extensive intervention. Major complications involve more severe cases, such as wound dehiscence greater than 2 cm and infections requiring surgical debridement.
  These secondary objectives are intended to assess the effect of preoperative nutritional optimization on postoperative recovery. The hypothesis is that improved nutritional status before surgery may result in fewer wound complications.

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared among researchers involved in the multicentric study across the hospitals of Delta Chirec, UZ Brussel, and Zuyderland Medical Center. This collaborative approach ensures that the research findings can be comprehensively analyzed and validated across multiple study sites, enhancing the overall quality and impact of the research.